CLINICAL TRIAL: NCT00931775
Title: Citalopram Versus Citalopram Plus Pindolol in Latency of Antidepressant Response Shortening in Major Depressive Disorder
Brief Title: Citalopram Versus Citalopram Plus Pindolol in Major Depressive Disorder
Acronym: CIT-PIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Enric Álvarez / Víctor Pérez, Hospital de la Santa Creu i Sant Pau. Psychiatry Department
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIT-PIN_01-0C3
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Major Depressive Disorder; Antidepressant Treatment Response
Keywords: Major depressive disorder, citalopram, pindolol, HDRS
MeSH Terms: conditions — Depressive Disorder, Major; Barakat syndrome | interventions — Pindolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citalopram + placebo (Placebo Comparator): Citalopram 20 mg/day t.i.d
  Interventions: Drug: Pindolol
- Citalopram + pindolol (Experimental): Citalopram 20 mg/day t.i.d Pindolol 15 mg/day t.i.d.
  Interventions: Drug: Pindolol

INTERVENTIONS:
Drug: Pindolol — Pill orally administered. 15 mg/day t.i.d.

SUMMARY:
The purpose of this study is to examine whether the speed of the clinical antidepressant action of citalopram can be accelerated by administering double doses of pindolol (15 mg/day, tid) which presumably should lead to increased 5-HT1A autoreceptor occupancy.

DETAILED DESCRIPTION:
Design, Settings, and Participants. A randomised, double-blind, placebo-controlled trial with MDD patients allocated to two treatment arms: citalopram + pindolol versus citalopram + placebo. Participants: outpatients with a depressive episode (DSM-IV criteria) were selected from a general hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a depressive episode
* HDRS score > 18
* Written informed consent

Exclusion Criteria:

* suicidal risk > 3
* severe organic illness
* other psychotropic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Scores on Hamilton Depression Rating Scale | 8 time points through 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enric Álvarez, MD, PhD, Principal Investigator — Department of Psychiatry. Hospital de la Santa Creu i Sant Pau; Víctor Pérez, MD, PhD, Study Director — Department of Psychiatry. Hospital de la Santa Creu i Sant Pau; Francesc Artigas, PhD, Study Chair — Neurochemistry department. Consejo Superior de Investigaciones Científicas
Locations (1):
- Outpatients Service of Psychiatry Department. Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Portella MJ, de Diego-Adelino J, Ballesteros J, Puigdemont D, Oller S, Santos B, Alvarez E, Artigas F, Perez V. Can we really accelerate and enhance the selective serotonin reuptake inhibitor antidepressant effect? A randomized clinical trial and a meta-analysis of pindolol in nonresistant depression. J Clin Psychiatry. 2011 Jul;72(7):962-9. doi: 10.4088/JCP.09m05827blu. Epub 2010 Oct 19. PMID 21034693